CLINICAL TRIAL: NCT06488859
Title: Affective Treatment Study
Brief Title: Affect Treatment for Depression and Anxiety (TAD Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Michelle Craske, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAD Pilot
Record Dates: First submitted 2024-06-24; First posted 2024-07-05 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Positive Affect Treatment (Experimental): 8 sessions of psychotherapy designed to augment reward anticipation, reward attainment, and reward learning.
  Interventions: Behavioral: Positive Affect Treatment
- Positive Affect Treatment and Negative Affect Treatment (Active Comparator): 8 sessions of psychotherapy. 3-5 sessions of psychotherapy designed to augment reward anticipation, reward attainment, and reward learning. Remaining sessions of psychotherapy designed to decrease threat avoidance, threat appraisal and arousal.
  Interventions: Behavioral: Positive Affect Treatment and Negative Affect Treatment

INTERVENTIONS:
Behavioral: Positive Affect Treatment — Sessions 1-8: Pleasurable activities + imaginal recounting and reinforcement of positive mood effects
  Arms: Positive Affect Treatment
Behavioral: Positive Affect Treatment and Negative Affect Treatment — Sessions 1-4: Pleasurable activities + imaginal recounting and reinforcement of positive mood effects Sessions 5-8: Exposure therapy to feared or avoided situations, sensations, or memories
  Arms: Positive Affect Treatment and Negative Affect Treatment

SUMMARY:
The goal of this study is to determine whether subjects who do not show expected clinical improvement during the early course of positive affect treatment (PAT) would benefit from switching to an alternative psychosocial treatment (negative affect treatment) that is designed to instead target and improve deficits in threat sensitivity.

Participants will complete laboratory tests, psychiatric assessments, and self-report questionnaires as part of the study.

The total length of participation is around 5 months.

DETAILED DESCRIPTION:
Anhedonia, or loss of interest or pleasure in usual activities, is characteristic of depression, some types of anxiety, as well as substance abuse and schizophrenia. Specifically, anhedonia is associated with deficits in the appetitive reward system. Previously, our team developed a novel transdiagnostic psychosocial treatment for anhedonia that was designed to specifically target and improve deficits in reward sensitivity: Positive Affect Treatment (PAT). In clinical trials, PAT has been proven to be clinically effective at increasing positive affect, reducing negative affect, and improving depression, anxiety and stress (Craske et al., 2019, Craske et al., 2023). Like all psychosocial interventions, however, PAT is not effective for every individual. The goal of the current study is to determine whether subjects who do not show expected clinical improvement during the early course of PAT would benefit from switching to an alternative psychosocial treatment (Negative Affect Treatment [NAT]) that is designed to instead target and improve deficits in threat sensitivity.

Upon enrollment, each participant will complete a two-week long baseline assessment period before beginning treatment. On the first day of the baseline period, participants will complete a brief anhedonia interview, which will be conducted by an independent interviewer over the phone or HIPAA-compliant Zoom. For this interview, participants will answer 3 items using a 4-point rating scale, which will then be rated by the interviewer. In addition, participants will complete a battery of psychosocial questionnaires (approx. 25 minutes) remotely via REDCap to assess their mood, current symptoms and impairment. The participant will complete this assessment (including the clinical interview and questionnaires) a total of four times throughout the study: (1) the first day of the baseline period, (2) just before their first treatment session (i.e., the last day of the baseline period), (3) at the point of switching to the second treatment stage, and (4) just after completing treatment. In addition, beginning on the first day of their baseline period and throughout the remainder of their participation, subjects will be asked to provide daily mood ratings using a 0-10 scale.

Following the baseline period, participants will receive weekly 60-minute individual therapy sessions remotely (via HIPAA-compliant Zoom) with a highly trained psychotherapist. Before each session, participants will complete a short (approx. 7-10 minutes) series of surveys/questions to monitor their symptoms and other important clinical changes.

All participants will receive a variation of the same treatment (PAT), however, participants who do not show the expected clinical improvement during the first 3-5 sessions of PAT will be switched to an alternative treatment (NAT). Participants who show clinical improvement in response to PAT will receive a total of 8 weeks of therapy. Participants who fail to show signs of clinical improvement in response to the first 3-5 sessions of PAT will discontinue PAT and begin NAT; they will receive a total of 8 weeks of therapy with NAT (in addition to the 3-5 weeks of therapy with PAT that they already completed).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Low positive affect indexed by less than or equal to 24 on the positive affect subscale of the PANAS (i.e., PANAS-P); and scores of greater than or equal to 11 for depression and greater to or equal to 6 for anxiety on the Depression, Anxiety, and Stress Scale.
* Score of greater than or equal to 4 on any WSAS subscale
* Willingness to refrain from starting other psychosocial or pharmacological treatments until study completion.

Exclusion Criteria:

* Patient report of serious medical conditions - such as history of serious, uncontrolled medical illness, or instability (including significant cardio-pulmonary disease, organic brain syndrome, seizure disorder, cerebrovascular disease, thyroid dysfunction, and diabetes)
* Current active suicidal ideation
* Lifetime history of bipolar disorder, psychosis, cognitive impairment, or organic brain damage
* Substance use disorder (including smoking) within the last 6 months. History of cocaine or stimulate use (e.g., amphetamine, cocaine, methamphetamine)
* Greater than 11 cigarettes per week or nicotine equivalent
* History of marijuana, cocaine or stimulant use 5-7 times/week or more before age 15 (e.g., amphetamine, cocaine, methamphetamine)
* Willingness to refrain from marijuana use 1 week before laboratory assessments
* Pregnancy
* Bupropion, dopaminergic or neuroleptic medications use in the past 6 months
* Heterocyclics and SSRIs are permitted if stabilized (3 months) and PRN benzodiazepines and beta-blockers are permitted but discouraged on laboratory assessment visits
* Refusal of video/audio-taping
* Prior participation in previous waves of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule Expanded (PANAS-X) (General Dimensions Scales) | Baseline (week 1), pre-treatment (week 2), mid-treatment (week 6), post-treatment (week 11/week 16, depending on treatment condition)
  Reported positive affect (general dimensions scale positive affect) and negative affect (general dimension scale negative affect) (score range for each scale: 10-50), higher scores represent higher levels of positive affect or negative affect).
Depression Anxiety and Stress Scale (DASS-21) | Baseline (week 1), pre-treatment (week 2), mid-treatment (week 6), post-treatment (week 11/week 16, depending on treatment condition)
  Reported symptoms of depression (score range: 0-21), anxiety (score range: 0-21), and stress (score range: 0-21), higher scores indicate higher severity and frequency.

SECONDARY OUTCOMES:
Interviewer Anhedonia Ratings | Baseline (week 1), pre-treatment (week 2), mid-treatment (week 6), post-treatment (week 11/week 16, depending on treatment condition)
  Interviewer ratings of interest, pleasure, and motivation in hobbies/pastimes, foods/drinks, social activities (score range: 1-12), higher scores indicate lower anhedonia
Behavioral Inhibition/Behavioral Activation (reward drive subscale) (BAS-RD) | Baseline (week 1), pre-treatment (week 2), mid-treatment (week 6), post-treatment (week 11/week 16, depending on treatment condition)
  Mediator: Reported reward sensitivity (score range: 4-16), and threat sensitivity (score range: 7-28), with higher scores indicating higher sensitivity
Beck Depression Inventory (BDI-9) | Baseline (week 1), pre-treatment (week 2), mid-treatment (week 6), post-treatment (week 11/week 16, depending on treatment condition)
  Reported suicidal ideation (score range: 0-3), higher scores indicate higher suicidality
Temporal Experience of Pleasure Scale (TEPS) | Baseline (week 1), pre-treatment (week 2), mid-treatment (week 6), post-treatment (week 11/week 16, depending on treatment condition)
  Change in reported anticipatory pleasure (score range: 10-60) and consummatory pleasure (score range: 8-48), higher scores indicate higher reward responsiveness
Dimensional Anhedonia Rating Scale (DARS) | Baseline (week 1), pre-treatment (week 2), mid-treatment (week 6), post-treatment (week 11/week 16, depending on treatment condition)
  Reported desire, motivation, effort, and consummatory pleasure across hedonic domains (score range: 0-104), higher scores indicate lower anhedonia
Work and Social Adjustment Scale (WSAS) | Baseline (week 1), pre-treatment (week 2), mid-treatment (week 6), post-treatment (week 11/week 16, depending on treatment condition)
  Reported impairment at work, home, and in relationships (score range: 0-40), higher scores indicate higher impairment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Southern Methodist University, Dallas, Texas